CLINICAL TRIAL: NCT04959370
Title: Comparison of Clinical Efficacy Between Dynamic Dip Screw and Cannulated Compression Screw for Fresh Femoral Neck Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PekingUTH ZF DHS
Record Dates: First submitted 2021-07-02; First posted 2021-07-13 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Femoral Neck Fractures
Keywords: Femoral neck fracture; Internal fixation of fracture; Dynamic hip screw; Cannulated compression screw
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Dynamic hip screw (DHS) (Experimental)
  Interventions: Device: internal fixation implantation of dynamic hip screw
- Cannulated compression screw (CCS) (Active Comparator)
  Interventions: Device: internal fixation implantation of cannulated compression screw

INTERVENTIONS:
Device: internal fixation implantation of dynamic hip screw — Dynamic hip screws (DHS) are a femoral head-sparing orthopedic device used to treat femoral neck fractures.
  Arms: Dynamic hip screw (DHS)
Device: internal fixation implantation of cannulated compression screw — Cannulated Screw is designed to provide a minimally invasive method of anatomical fixation.
  Arms: Cannulated compression screw (CCS)

SUMMARY:
For fresh femoral neck fracture internal fixation, both DHS and CCS can make strong fixation of hip and have good recovery. There is no statistical difference in complications after surgery between the two procedures. Patients with DHS internal fixation have earlier postoperative weight bearing, which is conducive to functional exercise of the injured limb. DHS internal fixation system is recommended for patients with unstable fractures and severe osteoporosis.

DETAILED DESCRIPTION:
Objective: To compare the clinical effect of dynamic hip screw (DHS) and cannulated compression screw (CCS) in the treatment of fresh femoral neck fracture. Methods: A retrospective study was conducted to analyze the data of 91 patients with fresh femoral neck fracture treated with DHS or CCS in our hospital from January 2012 to June 2016.The cases were divided into two groups according to internal fixation: 44 cases in the DHS group and 47 cases in the CCS group. By comparing operative time, intraoperative bleeding, postoperative load, Harris scoring and the complications such as postoperative necrosis of femoral head and shortening of femoral neck appearance, we evaluated the clinical curative effect of two kinds of fixation.

ELIGIBILITY:
Inclusion Criteria:

* fresh femoral neck fracture
* can walk before fracture
* less than 65 years old

Exclusion Criteria:

* Patients combined with other bone fractures.
* Pathological fracture (e.g., primary or metastatic tumor)
* Serious soft tissue injury, judged by the investigator, will impact the union of the fracture, combined open fractures, vascular injury, and combined osteofascial compartment syndrome.
* Multiple systemic injuries judged by researchers not suitable for enrollment. Revision surgeries (for example, due to malunion, nonunion or infection)
* Concurrent medical conditions judged by researchers not suitable for enrollment, such as: metabolic bone disease, post-polio syndrome, poor bone quality, prior history of poor fracture healing, etc
* Patients known to be allergic to implant components
* Patients who are currently using chemotherapeutics or accepting radiotherapy, use systematically corticosteroid hormone or growth factor, or long-term use sedative hypnotics (continuous use over 3 months) or non-steroidal anti-inflammatory drugs (continuous use over 3 months)
* Subjects have significant neurological or musculoskeletal disorders or may have adverse effects on gait or weight-bearing (e.g., muscular dystrophy, multiple sclerosis, cerebral infarction, hemiplegia, Charcot arthropathy, avascular necrosis of the femoral head).

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Internal fixation failure rate | from operation to 1-year follow-up after the surgery
  defined as the total incidence of internal plant cut-out and fracture.

SECONDARY OUTCOMES:
Number of Participants with Bone nonunion | from operation to 1-year follow-up after the surgery
  evaluate bone healing according to the lateral X-ray examination. According to the regulations of Food and Drug Administration of the US, if there are no obvious signs of fracture healing 9 months after the fracture, or if there is no obvious difference in fracture space after three consecutive months, it is defined as nonunion.
Harris hip score | from operation to 1-year follow-up after the surgery
  the score value is from 0 to 100, and a higher score means a better outcome
operation time | intraoperation
  from the incision to internal fixation implanted
The times of intraoperative fluoroscopy | intraoperation
  average 25 milliseconds per X-ray shot, record the number of X-ray shot
Number of Participants with Postoperative adverse events | from operation to 1-year follow-up after the surgery
  including ipsilateral femoral head avascular necrosis, infection, wound hematoma, ipsilateral coxa vara, and ipsilateral limb shortening
Garden index | from operation to 1-year follow-up after the surgery
  The fracture reduction will be considered unsatisfied if the index is less than 155 degrees or more than 180 degrees.
A 12-Item Short-Form Health Survey (SF-12) | from operation to 1-year follow-up after the surgery
  the score value is from 0 to 100, and a higher score means a better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China